CLINICAL TRIAL: NCT06500364
Title: Knotless Implants As an Alternative for Capsular Closure in Primary Hip Arthroscopy: a Prospective, Multi-Center Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: American Hip Institute (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIRR-01891
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Femoro Acetabular Impingement
Keywords: Hip arthroscopy; Hip capsule
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LoopLoc Arm (Experimental): The patients in this group will have the LoopLoc device used following their hip arthroscopy, to close the capsule.
  Interventions: Device: LoopLoc Arm
- Control Arm (Active Comparator): This is a control group, meaning they had their hip arthroscopy done without the use of the LoopLoc device.
  Interventions: Device: Control Arm

INTERVENTIONS:
Device: LoopLoc Arm — Patients in this intervention will have had a capsular closure performed using a LoopLoc device after their hip arthroscopy.
  Arms: LoopLoc Arm
Device: Control Arm — Patients in this intervention will have not had a capsular closure using a LoopLoc device after their hip arthroscopy.
  Arms: Control Arm

SUMMARY:
The purpose of this research is to see if the Arthrex LoopLocTM device is better for capsular closure during hip arthroscopy than other treatments available.

The hip capsule is the tissue that surrounds your hip joint. It stabilizes and supports your hip joint. During hip arthroscopy, this tissue must be cut through in order to perform the hip arthroscopy. Once the hip arthroscopy is completed, the surgeon might repair the capsule. Current ways of repairing the capsule include knotted suture that might irritate structures around the hip, leading to the possible formation of scar tissue and pain. The Arthrex LoopLocTM device is knotless and may lower the presence of irritation and scar tissue around the hip after surgery and might lead to better outcomes.

Therefore, researchers will compare patients who had the LoopLocTM device used to close their hip capsule during surgery to those who did not have the device used, to see if there is a difference in their outcomes following surgery.

DETAILED DESCRIPTION:
The purpose of the study is to perform a prospective multi-center study evaluating the feasibility of a knotless capsular closure device in patients undergoing primary hip arthroscopy.

All patients that meet study inclusion and exclusion criteria will then be informed about the study and given the IRB-approved consent form. All patients will learn about the study during a clinic visit and will have the opportunity to review the consent form and ask questions. All questions and concerns about study participation and the consent form will be addressed by staff and staff will ensure patient understanding of the consent form. The study participant will then sign and date the consent form, as well as the research staff obtaining consent. Consent can be withdrawn at any time the participant chooses either verbally or in writing.

Patients will be indicated by their physician for a capsular closuring using the LoopLocTM device. These patients will follow up for two years with their providers and researchers, who will collect their patient-reported and clinical outcomes. Data from this study will be analyzed to determine if the LoopLocTM device for capsular closure has better outcomes than the alternative treatments available.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary hip arthroscopy
* Patients younger than 60 years old.
* Patients who will receive capsular closure with the Arthrex LoopLocTM device following hip arthroscopy.

Exclusion Criteria:

* Patients that had previous hip surgery,
* Patients that had a center edge angle (CEA) less than 25 degrees or greater than 40 degrees.
* Patients that have a cartilage damage grade greater than or equal to 3.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Modified Harris Hip Score | 2 years
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome.

SECONDARY OUTCOMES:
Non-Arthritic Hip Score | 2 years
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome.
International Hip Outcome Tool | 2 years
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome.
Hip Outcome Score Sports-Specific Subscale | 2 years
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome.
Visual Analog Scale | 2 years
  Patient-reported outcome measure. Scale 0-10, 10 indicating most amount of pain possible.
Patient Satisfaction | 2 years
  Patient-reported outcome measure. Scale 0-10, 10 indicating the highest level of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- American Hip Institute Research Foundation, Des Plaines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barber FA, Lee Evanson JR. Editorial Commentary: Acetabular Labral Repair-Is A Knotless Anchor Better? Arthroscopy. 2019 Jan;35(1):77-79. doi: 10.1016/j.arthro.2018.09.003. PMID 30611369
- [Background] Carbone AD, Prabhavalkar O, Chishti Z, Curley AJ, Parsa A, Domb BG. Hip Capsular Repair Results in Improved Patient-Reported Outcomes and Survivorship: A Systematic Review of the Literature. Arthroscopy. 2023 Feb;39(2):488-497. doi: 10.1016/j.arthro.2022.11.013. Epub 2022 Nov 14. PMID 36395962
- [Background] Conaway WK, Martin SD. Puncture Capsulotomy During Hip Arthroscopy for Femoroacetabular Impingement: Preserving Anatomy and Biomechanics. Arthrosc Tech. 2017 Nov 27;6(6):e2265-e2269. doi: 10.1016/j.eats.2017.08.036. eCollection 2017 Dec. PMID 29349029
- [Background] Beck EC, Cvetanovich GL, Levy DM, Weber AE, Kuhns BD, Khair MM, Rasio J, Nho SJ. A T-capsulotomy provides increased hip joint visualization compared with an extended interportal capsulotomy: commentary response. J Hip Preserv Surg. 2019 Nov 23;6(3):290-291. doi: 10.1093/jhps/hnz043. eCollection 2019 Aug. No abstract available. PMID 31798933
- [Background] Domb BG, Chaharbakhshi EO, Perets I, Walsh JP, Yuen LC, Ashberg LJ. Patient-Reported Outcomes of Capsular Repair Versus Capsulotomy in Patients Undergoing Hip Arthroscopy: Minimum 5-Year Follow-up-A Matched Comparison Study. Arthroscopy. 2018 Mar;34(3):853-863.e1. doi: 10.1016/j.arthro.2017.10.019. Epub 2018 Jan 17. PMID 29373289
- [Background] Economopoulos KJ, Chhabra A, Kweon C. Prospective Randomized Comparison of Capsular Management Techniques During Hip Arthroscopy. Am J Sports Med. 2020 Feb;48(2):395-402. doi: 10.1177/0363546519894301. Epub 2019 Dec 31. PMID 31891553
- [Background] Looney AM, McCann JA, Connolly PT, Comfort SM, Curley AJ, Postma WF. Routine Capsular Closure With Hip Arthroscopic Surgery Results in Superior Outcomes: A Systematic Review and Meta-analysis. Am J Sports Med. 2022 Jun;50(7):2007-2022. doi: 10.1177/03635465211023508. Epub 2021 Aug 17. PMID 34403279
- [Background] Monroe EJ, Chambers CC, Zhang AL. Periportal Capsulotomy: A Technique for Limited Violation of the Hip Capsule During Arthroscopy for Femoroacetabular Impingement. Arthrosc Tech. 2019 Jan 28;8(2):e205-e208. doi: 10.1016/j.eats.2018.10.015. eCollection 2019 Feb. PMID 30906690
- [Background] Ortiz-Declet V, Mu B, Chen AW, Litrenta J, Perets I, Yuen LC, Domb BG. Should the Capsule Be Repaired or Plicated After Hip Arthroscopy for Labral Tears Associated With Femoroacetabular Impingement or Instability? A Systematic Review. Arthroscopy. 2018 Jan;34(1):303-318. doi: 10.1016/j.arthro.2017.06.030. Epub 2017 Aug 31. PMID 28866345
- [Background] Radha S, Hutt J, Lall A, Domb B, Lynch TS, Griffin D, Field RE, Chuck-Cakic J. Best practice guidelines for arthroscopic intervention in femoroacetabular impingement syndrome: results from an International Delphi Consensus Project-Phase 1. J Hip Preserv Surg. 2019 Dec 16;6(4):326-338. doi: 10.1093/jhps/hnz055. eCollection 2019 Dec. PMID 32015889
- [Background] Willimon SC, Briggs KK, Philippon MJ. Intra-articular adhesions following hip arthroscopy: a risk factor analysis. Knee Surg Sports Traumatol Arthrosc. 2014 Apr;22(4):822-5. doi: 10.1007/s00167-013-2728-0. Epub 2013 Oct 26. PMID 24162717